CLINICAL TRIAL: NCT02690285
Title: A Pilot Study of Rapid Haplotyping Procedure for Personalized Dosing of Dichloroacetate (DCA) in Healthy Volunteers Part 1: Rapid Haplotyping Procedure for Determining the Response of Patients to DCA. Part 2: Personalized Dosing of Dichloroacetate for the Treatment of Rare and Common Diseases
Brief Title: A Pilot Study of Rapid Haplotyping Procedure for Personalized Dosing of Dichloroacetate (DCA) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medosome Biotec LLC (Industry); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB201500995 - N; R43FD005349 (FDA); OCR15997 (Other: Universiy of Florida)
Record Dates: First submitted 2016-02-09; First posted 2016-02-24 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dichloroacetic Acid; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: glutathione transferase zeta 1 (GSTZ1) haplotyping (Other): The participants will have blood collection and cheek cell collection after signing the informed consent, to determine GSTZ1 haplotype.
  Interventions: Other: GSTZ1 haplotyping
- Part 2: Dichloroacetate (DCA) Kinetics (Experimental): Eight study participants will be administered oral Dichloroacetate (DCA) 25 mg/kg daily for 5 days. On the fifth day frequent blood samples will be obtain over the following 24 hours. Study participants will complete a DCA kinetic study on day 5, at the Clinical Research Clinic (CRC).
  Interventions: Drug: Dichloroacetate (DCA); Other: GSTZ1 haplotyping

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Dichloroacetate (DCA) 25 mg/kg oral solution will be administered daily for 5 days.
  Arms: Part 2: Dichloroacetate (DCA) Kinetics
Other: GSTZ1 haplotyping — One teaspoon of blood is collected by standard phlebotomy. Cheek cells are collected by standard brushing. Samples will be analyzed at two independent laboratories to validate methods for GSTZ1 haplotype analysis.
  Other Names: Blood collection; Cheek cell collection

SUMMARY:
The purpose of this study is to identify and analyze the frequency of GSTZ1 haplotypes in a healthy adult population and determine the pharmacokinetics of Dichloroacetate (DCA) metabolism based on haplotype analysis.

The DCA drug is the first targeted treatment for Pyruvate Dehydrogenase Complex Deficiency (PDCD).

This pilot study, focuses on developing a high throughput, sensitive and accurate screening test for determining glutathione transferase zeta 1 (GSTZ1) haplotype status in individuals who would be treated with DCA.

DETAILED DESCRIPTION:
Pyruvate dehydrogenase complex (PDC) deficiency (PDCD) is a rare disease of mitochondrial energy failure with the life of expectancy of affected children severely truncated. Treatment of PDCD remains a serious, unmet challenge. Dichloroacetate (DCA) represents the first targeted therapy for PDCD by stimulating residual PDC activity. Cumulative experience with DCA has revealed dose accumulation in a subset of the population. This can be abated through personalized dosing of DCA, assigned by haplotype variation in the gene encoding glutathione transferase zeta 1 (GSTZ1), which biotransforms DCA to glyoxylate. Haplotype variations in GSTZ1 influence the kinetics and dynamics of chronically administered DCA. A single dose of DCA has a bioavailability approaching unity and is widely distributed throughout the body. The plasma half-life (t ½) is ~1 hr in drug-naïve subjects. Gender does not influence DCA kinetics or metabolism. The major route of biotransformation is via dehalogenation to glyoxylate by glutathione transferase zeta 1 (GSTZ1). DCA is a mechanism-based inhibitor of GSTZ1, so repeated administration results in increased plasma t ½ and decreased clearance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as outline in the physical exam and blood tests
* Non smoker

Exclusion Criteria:

* Cannot comprehend or refuse to sign the informed consent form;
* Febrile or have other clinical signs of infection;
* Pregnant or are nursing;
* In females, cannot or refuse to use contraception or avoid unprotected intercourse during the study;
* Uncontrolled hypertension (BPs > 160 mmHg or BPd > 100 mmHg) on conventional medication;
* Anemic (hematocrit < 35% in males; < 35% in females;
* Serum creatinine ≥ 1.3 mg/dl, TSH > 4.5 mIU/ml; a transaminase (ALT or AST) > 2 x ULN, total bilirubin > 1.2 mg/dl or fasting glucose ≥ 110 mg/dl.
* History of psychosis, seizures or diabetes mellitus or be receiving anti-psychotic, anti-epileptic or blood glucose-lowering medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
GSTZ1 haplotype frequency | Baseline Visit
  The TagMan-based genotyping technology will be used for GSTZ1 haplotype analysis from both blood and cheek samples. Haplotype variations in GSTZ1 influence the kinetics of chronically administered investigational medication DCA. The coding region of the GSTZ1 gene contains three functionally important non-synonymous single nucleotide polymorphisms (SNPs) that give rise to five major GSTZ1 haplotypes: KRT (Z1A), KGT (Z1B), EGT (Z1C), EGM (Z1D), and KGM (Z1F).

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Dichloroacetate (DCA) | -10, 0, 5, 10, 20, 30 minutes and at 1, 2, 4, 6, 8, 12, 24, 30 hours post dose
  After 5 days of oral DCA administration, blood samples will be collected at the specified times for Peak Plasma Concentration (Cmax) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health: Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No